CLINICAL TRIAL: NCT06288646
Title: Using Infrared Spectroscopy to Analyze Volatile Organic Compounds (VOCs) in the Breath of Patients With Lung Cancer
Status: Terminated | Type: Observational
Why Stopped: Change in sponsor's business strategy (disease focus changed to breast cancer)
Sponsor: Breathe BioMedical Inc (Industry)
Collaborators: Vitalite Health Network (Unknown)
Responsible Party: Sponsor
Other Study IDs: ROMEO 101712
Record Dates: First submitted 2023-11-15; First posted 2024-03-01 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Lung Cancer; Non Small Cell Lung Cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Exhaled alveolar breath collected via a proprietary breath sampler
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Confirmed Lung Cancer: To be eligible for the lung cancer group:
  * Aged 50 and over;
  * Current or former smoker with smoking history ≥ 20 pack-years;
  * Capacity to give informed consent;
  * Non-metastatic non-small cell lung cancer, that has not been treated
  * No history of active cancer in the past 5 years (exceptions include: Ductal carcinoma in situ (DCIS), cervical intraepithelial neoplasia (CIN), non-invasive bladder cancer, non-melanoma skin cancers, Gleason prostate cancer ≤ 6);
  * Able to provide a breath sample.
  To be eligible for a second breath sample:
  * Same as above, in addition to, and with the exception of criterion 4:
  * Non-metastatic non-small cell lung cancer, which has undergone surgical resection;
  * 6 months since completion of surgery, radiation, and chemotherapy on primary NSCLC;
  * CT scan at least 6 months after surgical resection, confirming the absence of lung cancer.
- Control: For a participant to be eligible in the study control group:
  * Aged 50 and over;
  * Current or former smoker with smoking history ≥ 20 pack-years;
  * Capacity to give informed consent;
  * No history of active lung cancer;
  * No pulmonary nodule(s);
  * No active cancer in the last 5 years; (Note: DCIS, CIN, non-invasive bladder cancer, non-melanoma skin cancers, Gleason ≤ 6 prostate cancer will be exceptions);
  * Ability to provide a breath sample.
- Stable pulmonary nodule: For a participant to be eligible for admission to the stable lung nodules group:
  * Aged 50 and over;
  * Current or former smoker with smoking history ≥ 20 pack-years;
  * Capacity to give informed consent;
  * No history of active lung cancer or other active cancer in the past 5 years; (Note: DCIS, CIN, non-invasive bladder cancer, non-melanoma skin cancers, Gleason prostate cancer ≤ 6 or lower will be exceptions);
  * Presence of one or more stable lung nodules (as determined by the principal investigator);
  * Ability to provide a breath sample.

SUMMARY:
The goal of this clinical trial is to compare breath samples from patients with lung cancer, those with stable lung nodules, and individuals without lung cancer. The main questions it aims to answer are whether breath patterns are different in these groups and to see if breath patterns change after treatment in patients with lung cancer.

Participants will be asked to provide one breath sample, and two if they get treated. They will also be asked to fill out a questionnaire about their background and medical history.

DETAILED DESCRIPTION:
Globally, lung cancer accounts for the most cancer deaths in both sexes combined. It is believed to develop slowly through progressive accumulation of genetic mutations, hence the disease allows time for diagnosis and curative surgical treatment. Five year survival rates for non-small-cell lung carcinoma (NSCLC) can range from 57-61% when detected in the early stages of disease. This is compared with a survival rate of approximately 6% once distant metastases are present. However, disease diagnosis typically occurs when it has progressed to an advanced stage when patients present with signs and symptoms. Therefore, technologies capable of asymptomatic disease detection will significantly impact lung cancer specific mortality. Metabolomic profiling of cancer measures compounds produced as a result of cellular activity including volatile organic compounds (VOCs) in exhaled breath. Infrared spectroscopy is a proven technique for breath analysis that can measure chemical concentrations in the parts per trillion range for certain VOCs. When coupled with machine learning techniques, this has the potential to be a novel approach for disease detection using exhaled breath.

ELIGIBILITY:
Inclusion Criteria:

Study participants in the lung cancer and control cohorts must meet lung cancer screening criteria as defined by the PLCOm2012 and/or US Preventative Services Task Force (USPSTF) risk criteria.

Exclusion Criteria:

* Patients are not eligible if they are currently receiving treatment for lung cancer.
* Patients are not eligible for a second breath sample if it has been less than 6 months since last application of treatment.

Note: Breath sampling technology is sensitive to chemicals produced by tobacco, cannabis and e-cigarettes as well as alcohol (consumed by the subject or used by the operator around the equipment). We ask participants to refrain from:

* Smoking (tobacco, cannabis or e-cigarettes) at least 4 hours before breath sampling;
* Consume alcohol (including mouthwash) at least 8 hours before breath sampling.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants in all cohorts must meet lung cancer screening criteria as defined by the PLCOm2012 and/or US Preventative Services Task Force (USPSTF) risk criteria. This study will enroll 30 patients from 3 different cohorts (confirmed NSCLS, stable pulmonary nodules, screened and negative controls). Additionally, a second breath sample may be taken from the 30 patients with lung cancer, totalling up to 120 breath samples.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2023-04-24 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Differences in Breath Spectra of Lung Cancer, Stable Pulmonary Nodules, and Controls | 2 years
  Using infrared cavity-ringdown spectroscopy, breath spectra of volatile organic compounds (VOCs) will be measured. Breath spectra will be statistically analyzed to identify features specific to each of the respective cohorts. These features will be used to train mathematical and statistical models to differentiate and categorize the samples within the three cohorts.

SECONDARY OUTCOMES:
Differences in breath spectra of patients with lung cancer before and after treatment | 2 years
  Using infrared cavity ring-down spectrometry, breath samples will be taken from individual patients before and after surgical resection of the tumour. The objective is to identify and measure intra-patient differences in respiratory profiles before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Nada Hammami, Study Director — Vitalite Health Network; Marcel Mallet, MD, Principal Investigator — Vitalite Health Network
Locations (1):
- Vitalite Health Network, Moncton, New Brunswick, Canada